CLINICAL TRIAL: NCT00140998
Title: Estrogen Replacement in Hypogonadal Girls Treated With GH: Differential Effects of Mode of Estrogen Delivery
Brief Title: Estrogen Treatment (Oral vs. Patches) in Turner Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00-136
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-08

CONDITIONS: Turner Syndrome; Hypogonadism; Premature Ovarian Failure
Keywords: Turner syndrome; Hypogonadism; GH; Estrogen; Estrogen Patches; IGF-I; Body Composition; Protein Metabolism; Lipolysis
MeSH Terms: conditions — Turner Syndrome; Hypogonadism; Primary Ovarian Insufficiency | interventions — Estradiol

INTERVENTIONS:
Drug: 17 beta estradiol

SUMMARY:
The study attempts to evaluate if the way of administering estrogen, the principal female hormone, via patches or orally, affects the way estrogen works in girls with Turner Syndrome. These are girls who are very short and whose ovaries do not work. We will examine changes bone, protein and fat metabolism under the influence of estrogen delivered by a patch trough the skin vs estrogen taken orally. These studies are conducted while the girls are taking GH therapy.

DETAILED DESCRIPTION:
Girls with Turner Syndrome, between the ages of 10-16 years, were chosen as the study population. The study requires 3 overnight admissions to an in-patient Clinical Research Center(CRC). A baseline study is performed using stable isotope tracers of leucine, glycerol and glucose and serial blood sampling to measure protein and fat metabolism. Indirect calorimetry is used to measure substrate oxidation rates and total energy expenditure. DEXA scan is used to measure bone mineral density and body composition. Once the baseline study is complete subjects are randomly assigned to receive either estrogen orally or through a patch placed onto the skin in increasing doses changed every 2 weeks. After 6 weeks of estrogen treatment a second metabolic study, identical to the first, is performed, followed by a wash out period of 4 weeks. Subsequently, the subjects are switched to the alternate form of estrogen. At the end of 6 weeks a third and final metabolic study is repeated. All subjects continue to be on growth hormone throughout the study procedures.

ELIGIBILITY:
Inclusion Criteria:Girls with Turner syndrome 10-16 years old who are receiving growth hormone treatment.

-

Exclusion Criteria:Systemic disease or concomitant treatment wtih Oxandrolone. Significant obesity or chronic steroid use.

-

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16
Dates: Start 2001-01; Study Completion 2004-06

PRIMARY OUTCOMES:
Body Composition
Rates of whole body protein kinetics
Rates of whole body lipolysis

SECONDARY OUTCOMES:
Changes in IGF-I concentrations
Changes in Plasma Lipids

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States